CLINICAL TRIAL: NCT02496663
Title: A Phase I Trial of Osimertinib (AZD9291) and Necitumumab in EGFR-Mutant Non-Small Cell Lung Cancer After Progression on a Previous EGFR Tyrosine Kinase Inhibitor
Brief Title: Osimertinib and Necitumumab in Treating Patients With EGFR-Mutant Stage IV or Recurrent Non-small Cell Lung Cancer Who Have Progressed on a Previous EGFR Tyrosine Kinase Inhibitor
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01053; NCI-2015-01053 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-77; 9898 (Other: City of Hope Comprehensive Cancer Center LAO); 9898 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; necitumumab; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (osimertinib, necitumumab) (Experimental): Patients receive osimertinib PO QD on days 1-21 and necitumumab IV over 60 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA and CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Elastography; Procedure: Multigated Acquisition Scan; Biological: Necitumumab; Drug: Osimertinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Elastography — Undergo MRI
  Other Names: MRE
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Necitumumab — Given IV
  Other Names: Anti-Epidermal Growth Factor Receptor Monoclonal Antibody IMC-11F8; IMC 11F8; IMC-11F8; IMC11F8; Portrazza
Drug: Osimertinib — Given PO
  Other Names: AZD 9291; AZD-9291; AZD9291; Mereletinib

SUMMARY:
This phase I trial studies the safety, side effects and best dose of necitumumab when given together with osimertinib in treating patients with EGFR-mutant non-small cell lung cancer that is stage IV or has come back after a period of improvement (recurrent) and who have progressed on a previous EGFR tyrosine kinase inhibitor. Immunotherapy with monoclonal antibodies, such as necitumumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Osimertinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving necitumumab with osimertinib may be safe, tolerable in treating patients with EGFR-mutant non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of osimertinib (AZD9291) in combination with necitumumab in patients with EGFR-mutant non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVE:

I. To observe and record anti-tumor activity in these NSCLC patients in select cohorts of patients with EGFR-activating mutations including EGFR Exon 20 insertion mutations.

TRANSLATIONAL OBJECTIVES:

I. To characterize the pharmacokinetics of osimertinib (AZD9291) in combination with necitumumab.

II. To explore biomarkers of response and resistance to previous EGFR-tyrosine kinase inhibitors (TKIs) and with the combination by studying biopsied tumor tissue at baseline and at progression, as well as serial plasma deoxyribonucleic acid (DNA) specimens.

III. To create patient derived xenograft (PDX) models of patients with EGFR-mutant NSCLC both prior to study initiation and at acquired resistance to treatment.

OUTLINE: This is a dose-escalation study of necitumumab.

Patients receive osimertinib orally (PO) once daily (QD) on days 1-21 and necitumumab intravenously (IV) over 60 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) or multigated acquisition scans (MUGA) and computed tomography (CT) scan, magnetic resonance imaging (MRI) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 4 weeks, 8 weeks, every 12 weeks for 1 year, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV or recurrent/metastatic histologically confirmed non-small cell lung cancer (NSCLC)
* NSCLC must harbor at least one of the following EGFR activating mutations: Exon 21 L858R, Exon 19 deletion, Exon 18 G719X, Exon 21 L861Q or for EGFR Exon 20 insertion expansion cohort D, NSCLC must harbor an EGFR Exon 20 insertion performed by a Clinical Laboratory Improvement Act (CLIA) certified test
* For Dose escalation cohort - progressive disease on at least one prior EGFR-TKI (previous treatment with 3rd generation EGFR-TKI including osimertinib [AZD9291] allowed for dose escalation)
* For Dose Expansion Cohort A: patient must 1) have progression of disease on erlotinib, gefitinib or afatinib as last previous systemic treatment, 2) have biopsy of tumor taken after progression on erlotinib, gefitinib or afatinib which must be EGFR-T790M negative confirmed by central testing prior to treatment (if EGFR-T790M status is unknown, patients may consent for trial and for biopsy and testing for EGFR T790M will be performed as part of initial biopsy for trial), and 3) be treatment naive to 3rd generation EGFR-TKI (rociletinib, EGFR inhibitor HM61713 [HM61713] and osimertinib [AZD9291]) and EGFR monoclonal antibodies
* For Dose Expansion Cohort B (closed to accrual as of 8/30/18): patient must 1) have progression of disease on a 3rd generation EGFR-TKI such as AZD9291, rociletinib, HM61713, 2) be treatment naive to an EGFR monoclonal antibody, and 3) have a biopsy of tumor taken after progression on last EGFR-TKI that indicates loss of EGFR-T790M (EGFR-T790M negative) confirmed by central testing prior to treatment (if EGFR-T790M status is unknown, patients may consent for trial and for biopsy, and testing for EGFR T790M will be performed as part of initial biopsy for trial)
* For Dose Expansion Cohort C: patient must 1) have progression of disease on a 3rd generation EGFR-TKI such as osimertinib (AZD9291), rociletinib, HM61713, 2) be treatment naive to an EGFR monoclonal antibody, 3) have a biopsy of tumor taken after progression on last EGFR-TKI that indicates preservation of EGFR-T790M post-progression on 3rd generation EGFR-TKI with biopsy confirmation by central testing prior to treatment (if EGFR-T790M status is unknown, patients may consent for trial and for biopsy, and testing for EGFR T790M will be performed as part of initial biopsy for trial)
* For Dose Expansion Cohort D: patient must 1) tumor that harbors an EGFR Exon 20 insertion by a CLIA certified test, and 2) have progressive disease on or after platinum based chemotherapy, and 3) be treatment naïve to 3rd generation and beyond EGFR-TKI (i.e., osimertinib [AZD9291], poziotinib, TAK-778) and EGFR monoclonal antibody; patient who received 1st or 2nd generation EGFR-TKI (such as erlotinib, gefitinib, afatinib) are eligible provided that they did not achieve a response to treatment or they did not have a duration of treatment on EGFR-TKI of 6 months or more
* For Dose Expansion Cohort E: patient must have progressive disease on osimertinib (AZD9291) as first-line EGFR-TKI treatment for metastatic NSCLC; patients must also be treatment naive to EGFR-monoclonal antibody
* Adequate archival tissue from a biopsy performed after progression of disease on previous EGFR-TKI or willing to consent for a fresh tumor biopsy; (mandatory for Cohorts A, B, C; optional for dose escalation and Cohort D, and Cohort E)
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, defined as at least one lesion that can be accurately measured in at least one dimension >= 10 mm (>= 1 cm) by computed tomography (CT) imaging or magnetic resonance imaging (MRI) within 42 days prior to registration; the CT from a combined positron emission tomography (PET)/CT may be used only if it is of diagnostic quality; laboratory parameters are not acceptable as the only evidence of disease
* Any number of prior therapies is allowed
* Age >= 18 years. NSCLC is exceedingly rare in patients < 18 years of age. Because no dosing or adverse event data are currently available on the use of and necitumumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Patients must have the ability to swallow tablets
* Life expectancy of greater 3 months
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (patients with Gilbert's syndrome may have serum bilirubin > 1.5 ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal
* Creatinine =< 1.5 x ULN OR
* Creatinine clearance >= 50 mL/min
* The effects of osimertinib (AZD9291) and necitumumab on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception using one of the methods listed below prior to study entry, for the duration of study participation, and for 3 months for women and 6 months for men following the date of the last dose of osimertinib (AZD9291) and/or necitumumab:

  * Total abstinence from sexual intercourse (minimum one complete menstrual cycle prior to study drug administration);
  * Vasectomized male subject or vasectomized partner of female subjects
  * Hormonal contraceptives (oral, parenteral, transdermal or vaginal ring) prior to study drug administration; if the subject is currently using a hormonal contraceptive, she should also use a barrier method during this study and for 3 months after study completion;
  * Intrauterine device (IUD);
  * Double-barrier method: male condom plus diaphragm or vaginal cap with spermicide (contraceptive sponge, jellies or creams)
  * Additionally, for all methods above (except for abstinence), male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must use condoms for the duration of the study and for 6 months following completion of therapy
* Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to initiation of treatment; women will be considered not of childbearing potential if they are surgically sterile (bilateral oophorectomy or hysterectomy) and/or post menopausal (amenorrheic for at least 12 months); should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patients with untreated brain metastases are allowed provided that the patient is clinically asymptomatic and stable; patients with a prior history of symptomatic brain metastases are eligible provided:

  * The brain metastases have been treated
  * The patient is asymptomatic from the brain metastases at enrollment
  * Corticosteroids prescribed for the management of brain metastases have been discontinued at least 7 days prior to registration
  * The brain metastases are stable on pre-registration imaging
* Patients must have completed last chemotherapy >= 3 weeks or radiotherapy >= 2 weeks prior to receiving study drugs
* Patients must have recovered from adverse events attributable to previous treatment to =< grade 1, except for alopecia and sensory neuropathy =< grade 2
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Major surgery within 21 days of starting protocol treatment
* Patients must discontinue previous EGFR-TKI at least 7 days prior to study enrollment with the exception that patients on osimertinib (AZD9291) for cohorts B, C and E can continue osimertinib (AZD9291) and need not discontinue prior to enrollment
* Patients who are receiving any other investigational agents; patients must have discontinued any other investigational agents for at least 5 half-lives or 3 months, whichever is greater, prior to initiation of osimertinib (AZD9291) in an investigational setting
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 weeks prior); all patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects of CYP3A4
* Patients with active malignancies other than NSCLC or prior curatively treated malignancy at high risk of relapse during the study period with the exception of localized squamous or basal cell skin cancers
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, gastrointestinal disease limiting absorption of osimertinib (AZD9291) such as a malabsorption syndrome or inflammatory bowel disease or psychiatric illness/social situations that would limit compliance with study requirements
* Mean resting corrected QT interval (QTc using Fridericia's formula [QTcF]) > 470 msec
* Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiography (ECG) (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause torsades de pointes
* Left ventricular ejection fraction < 50% on echocardiogram or multi-gated acquisition (MUGA)
* The effects of osimertinib (AZD9291) and necitumumab on the developing human fetus are unknown; for this reason and because EGFR inhibitors are known to be teratogenic, pregnant women are excluded from this study; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother osimertinib (AZD9291) and necitumumab breastfeeding should be discontinued if the mother is treated with osimertinib (AZD9291) and necitumumab; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with osimertinib (AZD9291)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2016-05-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of necitumumab combined with osimertinib | 21 days
  Defined as the highest dose tested in which only 0 or 1 out of 6 evaluable patients experience a dose limiting toxicity, as graded by the National Cancer Institute (NCI) Common terminology Criteria for Adverse Events (CTCAE) version 5.0. The recommended phase II dose (RP2D) will be the MTD, pending review of other safety/tolerability considerations. The RP2D will be determined based upon the MTD in the dose escalation portion as well as other considerations such as toxicities at additional courses. After completing the 4 expansion cohorts, the dose level will be re-reviewed to confirm that the RP2D is in fact well tolerated.
Incidence of toxicity | Up to 1 year
  Will be graded according to NCI CTCAE version 5.0. Grade and attribution will be summarized by dose level, cycle, organ system and type.

SECONDARY OUTCOMES:
Objective response rate (ORR) in patients treated at the recommended phase II dose | Up to 1 year
  Will be graded according to Response Evaluation Criteria in Solid Tumors version 1.1. ORR will be calculated as the percent of patients in each of the expansion cohorts whose best confirmed response is complete response (CR) or partial response (PR). Point estimates and associated 90% confidence intervals will be calculated.
Progression-free survival (PFS) | From start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
  Kaplan-Meier plots will be used to summarize the progression-free survival. Medians and associated 95% confidence intervals will be calculated.
Disease control rate (DCR) with combination osimertinib and necitumumab | Up to 1 year
  DCR will be the proportion of patients in each of the expansion cohorts whose best confirmed response is CR, PR, or stable disease. Point estimates and associated 90% confidence intervals will be calculated.

OTHER OUTCOMES:
Pharmacokinetic (PK) parameters of osimertinib in combination with necitumumab | Prior to dosing on day 1 of course 2, 1, 2, 4, 6, 8, and 24 hours after dosing in course 2 (dose escalation and cohort A); prior to treatment on day 1 of course 2 for up to 4 courses (cohorts B, C, and D)
  The PK analyses will be descriptive and will permit comparison of the plasma levels of osimertinib and its metabolites in the presence of necitumumab (in this trial) with levels in other studies where osimertinib is given alone or combined with other drugs. We will estimate mean PK parameters as well as the between-patient variability. Results will be listed and plotted, by dose as well as by objective response, qualitative patterns will be described, and means and standard deviations will be calculated for use in planning follow-up studies.
Presence of biomarkers of response and resistance to previous EGFR-tyrosine kinase inhibitors | Up to 1 year
  Will study biopsied tumor tissue as well as serial plasma deoxyribonucleic acid specimens. For each cohort alone, Fisher's exact test, and in a stratified analysis including all cohorts, an exact logistic regression model, will be used to examine the association with objective response and a Cox proportional hazards model will be used to examine the association with PFS. Odds ratio's and hazard ratio's will be estimated and associated 90% two-sided confidence intervals will be constructed. Testing will be one-sided, at the 0.05-level.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Riess, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (15):
- United States (15):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Cancer Center Cary, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania